CLINICAL TRIAL: NCT01323816
Title: Process and Outcome Differences in Care Provided in Intensive Care Units (ICUs) With Physician Versus Nurse Practitioner First Responders
Brief Title: Differences in Care Provided in Intensive Care Units (ICUs) With Physician Versus Nurse Practitioner First Responders
Status: Completed | Type: Observational
Sponsor: Naeem Ali, MD (Other)
Responsible Party: Sponsor-Investigator, Naeem Ali, MD, Medical Director, Medical Intensive Care Unit (MICU);, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2009H0145
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Traditional: ICU staffed by a resident, pulmonary fellow and attending
  Interventions: Other: Medically directed care
- Non-Traditional: ICU staffed by Nurse Practitioners as the direct care deliverer, a pulmonary fellow, and an attending
  Interventions: Other: Medically directed care

INTERVENTIONS:
Other: Medically directed care — There is no research directed care. Patients are treated as medically indicated.

SUMMARY:
The purpose of this study is to evaluate and compare outcomes of patients that have received care in medical intensive care units in a tertiary care facility with two different models; the traditional model including resident, pulmonary fellow and attending physician and a nontraditional model which has Nurse Practitioners as the direct care deliverer, a pulmonary fellow, and an attending.

DETAILED DESCRIPTION:
This will be a retrospective cohort study that is performed between two medical intensive care units (ICU). The goal is to compare outcomes of patients that have received care in medical intensive care units in a tertiary care facility with two different models; the traditional model including a resident, pulmonary fellow and attending and a nontraditional model which has Nurse Practitioners as the direct care deliverer, a pulmonary fellow, and an attending. Outcomes that will be measured include ICU length of stay, hospital length of stay after ICU discharge, ventilator days, daily spontaneous breathing trials, and daily awakening trials, as well as mortality in hospital and after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to designated ICU between September 1, 2007 and September 30, 2010.

Exclusion Criteria:

* Not admitted to designated ICU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients being seen at designated ICU during the time period being investigated.
Sampling Method: Probability Sample
Enrollment: 3659 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Life-years hospital costs | 2007 - 2010
  Life-years per $10,000 hospital costs - defined as the sum of days of survival after ICU admission for all patients admitted to each ICU/sum of all hospital costs for all patients admitted to each ICU

SECONDARY OUTCOMES:
Intensive Care Unit (ICU) mortality | 2007 - 2010
Hospital mortality | 2007 - 2010
Time to death | 2007 - 2010
Ventilator Days | 2007 - 2010
Ventilator-free days | 2007 - 2010
  Days alive and not requiring mechanical ventilation in first 28 days after ICU admission
Intensive Care Unit (ICU)-free days | 2007 - 2010
  Days alive and not in the ICU in first 28 days after ICU admission
Evidence-based care | 2007 - 2010
  % of ICU days receiving evidence-based care will also be explored as mediators of other outcomes)
  * Sedation holidays
  * Spontaneous breathing trials
  * Days with continuous infusions of sedatives
  * Head of bed elevation
Discharge location among survivors | 2007 - 2010
Intensive Care Unit (ICU)Length of Stay (LOS) | 2007 - 2010
Hospital Length of Stay (LOS) | 2007 - 2010
Hospital costs | 2007 - 2010
Hospital charges | 2007 - 2010
Patient Satisfaction Survey Results | 2007 - 2010

CONTACTS AND LOCATIONS:
Overall Officials: Naeem Ali, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Cooper LM, Linde-Zwirble WT. Medicare intensive care unit use: analysis of incidence, cost, and payment. Crit Care Med. 2004 Nov;32(11):2247-53. doi: 10.1097/01.ccm.0000146301.47334.bd. PMID 15640637
- [Background] Halpern NA, Pastores SM, Greenstein RJ. Critical care medicine in the United States 1985-2000: an analysis of bed numbers, use, and costs. Crit Care Med. 2004 Jun;32(6):1254-9. doi: 10.1097/01.ccm.0000128577.31689.4c. PMID 15187502
- [Background] Kleinpell RM, Ely EW, Grabenkort R. Nurse practitioners and physician assistants in the intensive care unit: an evidence-based review. Crit Care Med. 2008 Oct;36(10):2888-97. doi: 10.1097/CCM.0b013e318186ba8c. PMID 18766097
- [Background] Mitchell-DiCenso A, Guyatt G, Marrin M, Goeree R, Willan A, Southwell D, Hewson S, Paes B, Rosenbaum P, Hunsberger M, Baumann A. A controlled trial of nurse practitioners in neonatal intensive care. Pediatrics. 1996 Dec;98(6 Pt 1):1143-8. PMID 8951267
- [Background] Pronovost PJ, Angus DC, Dorman T, Robinson KA, Dremsizov TT, Young TL. Physician staffing patterns and clinical outcomes in critically ill patients: a systematic review. JAMA. 2002 Nov 6;288(17):2151-62. doi: 10.1001/jama.288.17.2151. PMID 12413375
- [Background] Treggiari MM, Martin DP, Yanez ND, Caldwell E, Hudson LD, Rubenfeld GD. Effect of intensive care unit organizational model and structure on outcomes in patients with acute lung injury. Am J Respir Crit Care Med. 2007 Oct 1;176(7):685-90. doi: 10.1164/rccm.200701-165OC. Epub 2007 Jun 7. PMID 17556721